CLINICAL TRIAL: NCT04333953
Title: Prospective Observational Study for Patients With HIV and Confirmed SARS-CoV-2
Brief Title: COVID-19 in Patients With HIV
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Dima Dandachi, Assistant Professor of Clinical Medicine, University of Missouri-Columbia
Other Study IDs: 2021341
Record Dates: First submitted 2020-03-31; First posted 2020-04-03 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: HIV/AIDS; COVID-19; SARS-CoV-2
Keywords: HIV; AIDS; COVID-19; SARS-CoV-2; clinical presentation; progression; clinical outcome
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; COVID-19; Disease Progression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention, observational study

SUMMARY:
Currently, limited data is available about patients with HIV in the context of the COVID-19 pandemic. People with HIV who have not achieved viral suppression through antiretroviral treatment may have a compromised immune system that leaves them vulnerable to infections and disease progression. However, little is known about the presentation and clinical outcomes of patients with HIV and SARS-CoV-2.

Our aim is to characterize the clinical presentation and disease course of COVID-19 in patients with HIV.

DETAILED DESCRIPTION:
Currently, limited data is available about patients with HIV in the context of the COVID-19 pandemic. People with HIV (PWH)/AIDS, or people with HIV who have not achieved viral suppression through antiretroviral treatment may have at higher risk for SARS-CoV-2 infections and disease progression. At present there is no evidence to suggest that there is an increased risk of infection and increased severity of illness for PWH. We know that during the SARS and MERS outbreaks, there were only few case reports of mild disease among PWH. Current clinical data suggest the main mortality risk factors are linked to older age and other co-morbidities. However, some healthy people have also developed severe disease from the SARS-CoV-2 infection.

This is a multi-center prospective observational study. Our aim is to characterize the clinical presentation and clinical course of COVID-19 in patients with HIV.

Patients with HIV and confirmed SARS-Cov-2 will be identified during routine clinical care in the inpatient or outpatient setting.

Contributors will share de-identified demographic data, health history data, and clinical data pertaining the patient's presentation with COVID-19 and outcomes obtained during routine care for their patients, using the secure online data collection tool REDCap.

ELIGIBILITY:
Inclusion Criteria:

* HIV disease
* Laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) or other commercial or public health assay

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with HIV disease who are diagnosed with COVID-19, inpatient or outpatient
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  COVID-19 related death among patients with HIV and COVID-19

SECONDARY OUTCOMES:
Frequency of patients requiring hospital admissions | 30 days
  Percentage of patients who required hospitalization
Frequency of patients requiring ICU admissions | 30 days
  Percentage of patients who required ICU admission
Frequency of respiratory support use | 30 days
  Percentage of patients who required respiratory support (new oxygen use, non-invasive ventilation,or invasive ventilation)
Frequency of kidney injury | 30 days
  Percentage of patients who developed acute kidney injury defined as increase in baseline creatinine, or use of renal replacement therapy
Frequency of liver injury | 30 days
  Percentage of patients who developed liver injury defined as increase in baseline ALT

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dandachi D, Geiger G, Montgomery MW, Karmen-Tuohy S, Golzy M, Antar AAR, Llibre JM, Camazine M, Diaz-De Santiago A, Carlucci PM, Zacharioudakis IM, Rahimian J, Wanjalla CN, Slim J, Arinze F, Kratz AMP, Jones JL, Patel SM, Kitchell E, Francis A, Ray M, Koren DE, Baddley JW, Hill B, Sax PE, Chow J. Characteristics, Comorbidities, and Outcomes in a Multicenter Registry of Patients With Human Immunodeficiency Virus and Coronavirus Disease 2019. Clin Infect Dis. 2021 Oct 5;73(7):e1964-e1972. doi: 10.1093/cid/ciaa1339. PMID 32905581